CLINICAL TRIAL: NCT01813292
Title: Comparative Study of Fluoride Metabolism, Bone Remodelling and Mineral Density in HIV + Men Being Given Tenofovir With FTC, Emtricitabine (TRUVADA®), or Without (VIREAD®), as Part of Their Antiretroviral Therapy.
Brief Title: Fluoride Metabolism, Bone Remodelling and Mineral Density in HIV Patients Treated With Tenofovir +/- Emtricitabine
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Célia Lloret-Linares, MD PhD, Professor, Medicine A Department,, Hopital Lariboisière
Other Study IDs: URT-Bone-001
Record Dates: First submitted 2013-03-12; First posted 2013-03-18 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: HIV Seropositivity
Keywords: male patients; treated by TRUVADA® or VIREAD® for more than 60 months
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
HIV+ patients are considered at risk for excessive bone fragility. Several factors could contribute: age, male sex, low body mass index (BMI), HIV infection per se, vitamin D deficiency, using tenofovir/a protease inhibitor (time on and/or current use). Tenofovir is used in a backbone of nucleosides/nucleotides analogues with emtricitabine (FTC), licensed as TRUVADA®, or without this analogue, licensed as VIREAD®. FTC closely resembles lamivudine (3TC) but is 5-fluorinated, the daily intake of fluoride is ~15 mg. Fluoride induces bone formation by stimulating osteoblasts, of often impaired bone quality.

The aim of the study is to compare in a cross-sectional design fluoride levels, bone renewal, bone mineral density (BMD) in HIV+ male patients treated by TRUVADA® or VIREAD® for more than 60 months. The patients will be randomly selected, then matched according to age, ethnic origin, BMI.

DETAILED DESCRIPTION:
Fluoride metabolism will be studied by measurement of fluoride in blood and in daily urine, bone remodelling by measurement of P1NP. Dual X-ray absorptiometry (DXA) will be used to determine the areal bone mineral density (aBMD) of the lumbar spine, femoral neck and distal radius. Volumetric BMD (v-BMD) and micro-architecture of distal radius and tibia will be studied using a HR-pQCT scan (Xtreme, Scanco).

ELIGIBILITY:
Inclusion Criteria:

* HIV+ patients
* male patients
* patients treated by tenofovir+emtricitabine(TRUVADA®) or tenofovir(VIREAD®) for more than 60 months.

Exclusion Criteria:

* chronic use of fluoroquinolones, antifungal agents, steroids
* malignancy (current or previous) requiring chemotherapy or radiotherapy

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV+ male patients treated by TRUVADA® or VIREAD® for more than 60 months.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Areal bone mineral density (aBMD) of the lumbar spine, femoral neck and distal radius measured by Dual X-ray absorptiometry (DXA) | ongoing, during the study period, according to the availability of DXA

CONTACTS AND LOCATIONS:
Overall Officials: Pierre O Sellier, M.D, Ph.D, Principal Investigator — Hopital Lariboisiere, Paris, France
Locations (1):
- Hopital Lariboisiere, Paris, France

IPD SHARING:
Plan to Share IPD: No